CLINICAL TRIAL: NCT00978029
Title: A 28-Day Study Evaluating the Safety of Ragweed (Ambrosia Artemisiifolia) Sublingual Tablet (SCH 39641) in Adult Subjects 50 Years of Age and Older With Ragweed-Induced Rhinoconjunctivitis (Protocol No. P06081)
Brief Title: Safety Study of Ragweed Allergy Immunotherapy Tablet in Subjects 50 Years of Age and Older (Study P06081)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P06081; MK-3641-004 (Other: Merck)
Record Dates: First submitted 2009-09-11; First posted 2009-09-16 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Rhinoconjunctivitis; Rhinitis; Conjunctivitis; Allergy
Keywords: immunotherapy
MeSH Terms: conditions — Rhinitis; Conjunctivitis; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Matching placebo tablet sublingual, once daily
  Interventions: Drug: Placebo
- SCH 39641 6 Amb a 1-U (Experimental): 6 Units Short Ragweed (Ambrosia artemisiifolia) Major Allergen 1 (Amb a 1-U) in an AIT, sublingual, once daily
  Interventions: Biological: SCH 39641
- SCH 39641 12 Amb a 1-U (Experimental): 12 Amb a 1-U in an AIT, sublingual, once daily
  Interventions: Biological: SCH 39641

INTERVENTIONS:
Drug: Placebo — Placebo sublingual tablet, once daily
  Arms: Placebo
Biological: SCH 39641 — Allergy immunotherapy tablet (sublingual)
  Other Names: MK-3641
  Arms: SCH 39641 6 Amb a 1-U
Biological: SCH 39641 — Allergy immunotherapy tablet (sublingual)
  Other Names: MK-3641
  Arms: SCH 39641 12 Amb a 1-U

SUMMARY:
The purpose of this study was to assess the safety and tolerability of a ragweed allergy immunotherapy tablet (AIT) administered sublingually (under-the tongue) in subjects 50 years of age and older with ragweed-induced rhinoconjunctivitis, with or without asthma.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 50 years of age or older, of either sex, and of any race/ethnicity.
* Subject must have a clinical history of ragweed-induced allergic rhinoconjunctivitis with or without asthma.
* Subject must have a positive skin prick test response to Ambrosia artemisiifolia at the Screening Visit
* Subject must have a forced expiratory volume in 1 second (FEV1) of at least 70% of predicted value at the Screening Visit and at Randomization.
* A subject's clinical laboratory tests, electrocardiogram (ECG) and vital signs conducted at the Screening Visit must be within normal limits or clinically acceptable to the investigator.

Exclusion Criteria:

* Subject with asthma who requires inhaled corticosteroids for the treatment of their asthma during the study period.
* Subject requiring anti-allergy medications during the time period from randomization to study completion.
* Subject who has received an immunosuppressive treatment within 3 months prior to the Screening Visit (except steroids for allergic and asthma symptoms).
* Subject with a history of anaphylaxis with cardiorespiratory symptoms.
* Subject with a history of chronic urticaria or angioedema.
* Subject with current severe atopic dermatitis.
* Female subject who is breastfeeding, pregnant, or intending to become pregnant.
* Subject with a history of allergy, hypersensitivity or intolerance to the ingredients of the investigational medicinal products (IMPs) (except for Ambrosia artemisiifolia), or self-injectable epinephrine.
* Subject with a history of self-injectable epinephrine use.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

REFERENCES:
- [Derived] Nolte H, Amar N, Bernstein DI, Lanier BQ, Creticos P, Berman G, Kaur A, Hebert J, Maloney J. Safety and tolerability of a short ragweed sublingual immunotherapy tablet. Ann Allergy Asthma Immunol. 2014 Jul;113(1):93-100.e3. doi: 10.1016/j.anai.2014.04.018. Epub 2014 May 14. PMID 24836393

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to non-compliance with Good Clinical Practice (GCP) 7 randomized participants who completed treatment were excluded from all subsequent analysis.
Groups:
- SCH 39641 6 Amb a 1-U: 6 Units Short Ragweed (Ambrosia artemisiifolia) Major Allergen 1 (Amb a 1-U) in an Allergy Immunotherapy Tablet (AIT) sublingual, once daily
Period: Overall Study
Arm/Group | Placebo | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U
Started | 65 | 66 | 65
Completed | 64 | 63 | 59
Not Completed | 1 | 3 | 6
Not completed — Adverse Event | 1 | 2 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- SCH 39641 6 Amb a 1-U: 6 Amb a 1-U in an AIT, sublingual, once daily
- Total: Total of all reporting groups
Arm/Group | Placebo | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U | Total
Number analyzed (Participants) | 65 | 66 | 65 | 196
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.4 (4.7) | 56.4 (5.4) | 56.2 (5.7) | 56.3 (5.3)
Gender [Count of Participants; unit: Participants]
  Female | 38 | 43 | 40 | 121
  Male | 27 | 23 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants Reporting Treatment-emergent Adverse Events (AEs)
Description: Participants were treated for 28 days with either 6 or 12 Units of SCH 39641 or placebo, and the proportion with treatment-emergent AEs were recorded. An AE is any unfavorable and unintended sign, symptom or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. Treatment-emergent AEs are new AEs that occur after participants have been randomized into the trial, or existing AEs that occurred during Screening that increase in severity after randomization.
Time Frame: Up to Day 42
Population: All subjects as treated (ASAT) consisting of all randomized participants who received at least one dose of study treatment. Due to non-compliance with GCP 7 participants were excluded from this analysis.
Measure: Number; unit: Proportion of Participants
Arm/Group | Placebo | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U
Number analyzed (Participants) | 65 | 66 | 65
Proportion of Participants | 0.446 | 0.515 | 0.615
Statistical Analysis 1: Comparison: Placebo vs SCH 39641 6 Amb a 1-U; Test type: Superiority or Other; p = 0.486, Fisher Exact; Percent Difference = 6.9, 95% CI 2-sided [-10.17 to 23.97]
Statistical Analysis 2: Comparison: Placebo vs SCH 39641 12 Amb a 1-U; Test type: Superiority or Other; p = 0.078, Fisher Exact; Percent Difference = 16.9, 95% CI 2-sided [0.01 to 33.83]

2. Secondary Outcome: Proportion of Participants Reporting Oral Pruritus
Description: Participants were treated for 28 days with either 6 or 12 Units of SCH 39641 or placebo, and the proportion with oral pruritus were reported.
Time Frame: Up to Day 42
Population: ASAT consisting of all randomized participants who received at least one dose of study treatment. Due to non-compliance with GCP 7 participants were excluded from this analysis.
Measure: Number; unit: Proportion of Participants
Arm/Group | Placebo | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U
Number analyzed (Participants) | 65 | 66 | 65
Proportion of Participants | 0.015 | 0.167 | 0.169

3. Secondary Outcome: Proportion of Participants Reporting Ear Pruritus
Description: Participants were treated for 28 days with either 6 or 12 Units of SCH 39641 or placebo, and the proportion with ear pruritus were reported.
Time Frame: Up to Day 42
Population: as for outcome 2
Measure: Number; unit: Proportion of Participants
Arm/Group | Placebo | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U
Number analyzed (Participants) | 65 | 66 | 65
Proportion of Participants | 0 | 0.061 | 0.077

4. Secondary Outcome: Proportion of Participants Reporting Throat Irritation
Description: Participants were treated for 28 days with either 6 or 12 Units of SCH 39641 or placebo, and the proportion with throat irritation were reported.
Time Frame: Up to Day 42
Population: as for outcome 2
Measure: Number; unit: Proportion of Participants
Arm/Group | Placebo | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U
Number analyzed (Participants) | 65 | 66 | 65
Proportion of Participants | 0.015 | 0.121 | 0.077

5. Secondary Outcome: Proportion of Participants Reporting Mouth Oedema
Description: Participants were treated for 28 days with either 6 or 12 Units of SCH 39641 or placebo, and the proportion with mouth oedema were reported.
Time Frame: Up to Day 42
Population: as for outcome 2
Measure: Number; unit: Proportion of Participants
Arm/Group | Placebo | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U
Number analyzed (Participants) | 65 | 66 | 65
Proportion of Participants | 0 | 0.015 | 0

6. Secondary Outcome: Proportion of Participants Who Discontinued Due to Adverse Events.
Description: Participants were treated for 28 days with either 6 or 12 Units of SCH 39641 or placebo, and the proportion with AEs leading to study discontinuation were reported. An AE is any unfavorable and unintended sign, symptom or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Up to Day 28
Population: as for outcome 2
Measure: Number; unit: Proportion of Participants
Arm/Group | Placebo | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U
Number analyzed (Participants) | 65 | 66 | 65
Proportion of Participants | 0.015 | 0.03 | 0.077

ADVERSE EVENTS:
Time Frame: Up to Day 42
Description: ASAT consisting of all randomized participants who received at least one dose of study treatment. Due to non-compliance with GCP 7 participants were excluded from this analysis.
Arm/Group | Placebo | SCH 39641 6 Amb a 1-U | SCH 39641 12 Amb a 1-U
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/66 | 1/65
Other Adverse Events (participants affected / at risk) | 11/65 | 23/66 | 23/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=65) | SCH 39641 6 Amb a 1-U (N=66) | SCH 39641 12 Amb a 1-U (N=65)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=65) | SCH 39641 6 Amb a 1-U (N=66) | SCH 39641 12 Amb a 1-U (N=65)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 4 (5) | 5 (5)
Eye pruritus (Eye disorders) | 4 (4) | 2 (2) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (6)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (5)
Oral pruritus (Gastrointestinal disorders) | 1 (1) | 11 (15) | 11 (21)
Paraesthesia oral (Gastrointestinal disorders) | 3 (3) | 3 (3) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (11) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor for review 45 days prior to submission for publication or presentation, copies of abstracts or manuscripts for publication that report any results of the trial. If the parties disagree concerning the sponsor's confidential information, the investigator agrees to meet with the sponsor's representative, prior to submission for publication, in order to make good faith efforts to discuss and resolve any issues or disagreements.